CLINICAL TRIAL: NCT00443430
Title: Trial of Early Aggressive Therapy in Juvenile Idiopathic Arthritis (TREAT in JIA)
Brief Title: Trial of Early Aggressive Drug Therapy in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Amgen (Industry)
Responsible Party: Principal Investigator, Carol Wallace, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AR049762 (NIH); 5R01AR049762-02 (NIH)
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Juvenile Chronic Polyarthritis; Juvenile Idiopathic Arthritis; Juvenile Rheumatoid Arthritis
Keywords: Childhood Arthritis; Juvenile Arthritis; Juvenile Arthritis Treatment; Childhood Arthritis Drug Treatment; Juvenile Arthritis Remission; Inactive Disease in Juvenile Arthritis; Childhood Polyarthritis; Extended Oligoarthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Methotrexate; Etanercept; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate Arm (Active Comparator): Methotrexate 0.5 mg/kg given by subcutaneous injection once per week, plus placebo etanercept and placebo prednisolone
  Interventions: Drug: methotrexate
- Methotrexate-Etanercept-Prednisolone Arm (Active Comparator): Methotrexate 0.5 mg/kg given by subcutaneous injection once per week, plus etanercept 0.8 mg/kg given by subcutaneous injection once per week, plus prednisolone by mouth daily with decreasing dose tapered over 16 weeks
  Interventions: Drug: methotrexate - etanercept - prednisolone arm

INTERVENTIONS:
Drug: methotrexate — Methotrexate 0.5 mg/kg given by sub cutaneous injection once per week, plus placebo etanercept and and placebo prednisolone
  Other Names: placebo enbrel; placebo prednisolone
  Arms: Methotrexate Arm
Drug: methotrexate - etanercept - prednisolone arm — methotrexate 0.5 mg/kg given by sub cutaneous injection once per week, plus etanercept 0.8 mg/kg given by sub cutaneous injection once per week, plus prednisolone, by mouth daily with decreasing dose tapered over 16 weeks.
  Other Names: enbrel; prednisone
  Arms: Methotrexate-Etanercept-Prednisolone Arm

SUMMARY:
The purpose of this study is to compare two aggressive drug regimens for children with poly-juvenile idiopathic arthritis (JIA) and extended oligo JIA.

DETAILED DESCRIPTION:
JIA is a type of arthritis with no definite cause and an onset prior to 16 years of age. JIA causes joint destruction, pain, and permanent disability. There are multiple types of JIA; collectively, they represent one of the most common chronic diseases in children and the most prevalent pediatric rheumatic illness. Poly-JIA, one type of JIA, affects at least five joints in the body within the first 6 months of disease. Long-term remission of poly-JIA is uncommon, and most children must remain on multiple combinations of medications for many years. The usual treatment for poly-JIA is based upon the gradual addition of medications that might be more effective in treating this disease. There is a need to find uniformly effective treatments for children with poly-JIA. Based on previous adult arthritis studies, there appears to be an early window of opportunity in the disease progression during which aggressive therapy has a profound beneficial long-term effect. The purpose of this study is to compare the effectiveness of two aggressive drug regimens in treating children with poly-JIA. Specifically, the study will determine whether aggressive therapy started in the first 6 months of disease onset can result in inactive disease and clinical remission while on these medications.

All participants will receive weekly methotrexate shots while in the study. In addition, participants will be randomly assigned to one of two groups:

* Group 1 participants will receive placebo etanercept shots for up to 12 months and daily placebo prednisolone liquid for 4 months.
* Group 2 participants will receive etanercept shots for up to 12 months and daily prednisolone liquid for 4 months.

The study will last up to 12 months and include two parts. Part A will last 1 to 6 months, depending on response to assigned treatments. If participants are still experiencing active arthritis at 6 months, they will be offered open-label treatment with etanercept and prednisolone. If participants experience inactive disease any time prior to 6 months, they will enter Part B of the study. During Part B, which will last up to 6 months, participants will remain on the same treatment regimen that they were provided in Part A. If participants experience inactive disease followed by a flare of disease any time during the study, they will stop participating.

During the study, there will be 11 study visits for all participants. Study visits will include a physical exam, including joint evaluations; blood and urine collection; and questionnaires regarding function, quality of life, medication compliance, other medications used, infections, and adverse symptoms.

Blood will be collected for translational studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active poly-JIA as determined by International League of Associations for Rheumatology (ILAR) criteria
* Onset of signs and symptoms of poly-JIA for 12 months or less prior to study screening
* Willing to use acceptable forms of contraception for the duration of the study and for 3 months after the study
* Parent or guardian willing to provide informed consent
* Able to attend all study visits

Exclusion Criteria:

* Received or currently receiving disease-modifying antirheumatic drugs (DMARDs), biologic, or prednisone for any duration for treatment of poly-JIA, with the following exceptions:

  1. Methotrexate duration must be less than or equal to 6 weeks at a dose of less than or equal to 0.5 mg/kg/week (40 mg max),
  2. Steroid use has been less than or equal to 4 weeks and the subject is off of steroids for at least 1 week prior to enrollment
* Received intramuscular or soft-tissue injections of corticosteroids for treatment of poly-JIA before receiving the first dose of study medication. Up to 2 joint injections with intra-articular steroids (IAS) will be allowed up to 7 days after the baseline visit.
* History of or active cancer of any type
* Active gastrointestinal disease (e.g., inflammatory bowel disease)
* Chronic or acute kidney or liver disorder
* Significant blood clotting defect
* AST (SGOT), ALT (SGPT), or BUN levels more than two times the upper level of normal, creatinine levels more than 1.5 mg/dl, or any other laboratory abnormality considered to be clinically significant within 28 days prior to baseline
* Chronic condition (e.g., diabetes, epilepsy) that is either not stable or poorly controlled and may interfere with study participation
* Received any investigational medication within 30 days prior to the first dose of study medication or scheduled to receive an investigational drug (other than the study medications) during the course of the study
* Chronic or active infection or any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 30 days prior to study screening
* HIV infected
* Known past or current hepatitis infection
* Received a live virus vaccine within 1 month prior to baseline
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Pregnancy
* Any medical condition that would make study participation difficult or inadvisable in the opinion of the investigator
* History of or current psychiatric illness that would interfere with study participation
* History of alcohol or drug abuse within the 6 months prior to study entry that would interfere with study participation
* Inability to comply with study requirements for any reason

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Wallace, MD, Principal Investigator — Childrens Hospital and Regional Medical Center
Locations (15):
- United States (15):
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Children's Hospital of Boston, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Texas Scottish Rite Hospital, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Lovell DJ, Reiff A, Jones OY, Schneider R, Nocton J, Stein LD, Gedalia A, Ilowite NT, Wallace CA, Whitmore JB, White B, Giannini EH; Pediatric Rheumatology Collaborative Study Group. Long-term safety and efficacy of etanercept in children with polyarticular-course juvenile rheumatoid arthritis. Arthritis Rheum. 2006 Jun;54(6):1987-94. doi: 10.1002/art.21885. PMID 16732547
- [Background] Wallace CA. Current management of juvenile idiopathic arthritis. Best Pract Res Clin Rheumatol. 2006 Apr;20(2):279-300. doi: 10.1016/j.berh.2005.11.008. PMID 16546057
- [Background] Wallace CA, Ruperto N, Giannini E; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology International Trials Organization; Pediatric Rheumatology Collaborative Study Group. Preliminary criteria for clinical remission for select categories of juvenile idiopathic arthritis. J Rheumatol. 2004 Nov;31(11):2290-4. PMID 15517647
- [Derived] Lim LSH, Lokku A, Pullenayegum E, Ringold S. Probability of Response in the First Sixteen Weeks After Starting Biologics: An Analysis of Juvenile Idiopathic Arthritis Biologics Trials. Arthritis Care Res (Hoboken). 2023 Jun;75(6):1238-1249. doi: 10.1002/acr.25003. Epub 2023 Jan 18. PMID 36651601
- [Derived] Jiang K, Wong L, Sawle AD, Frank MB, Chen Y, Wallace CA, Jarvis JN. Whole blood expression profiling from the TREAT trial: insights for the pathogenesis of polyarticular juvenile idiopathic arthritis. Arthritis Res Ther. 2016 Jul 7;18(1):157. doi: 10.1186/s13075-016-1059-1. PMID 27388672
- [Derived] Wallace CA, Giannini EH, Spalding SJ, Hashkes PJ, O'Neil KM, Zeft AS, Szer IS, Ringold S, Brunner HI, Schanberg LE, Sundel RP, Milojevic DS, Punaro MG, Chira P, Gottlieb BS, Higgins GC, Ilowite NT, Kimura Y, Johnson A, Huang B, Lovell DJ; Childhood Arthritis and Rheumatology Research Alliance (CARRA). Clinically inactive disease in a cohort of children with new-onset polyarticular juvenile idiopathic arthritis treated with early aggressive therapy: time to achievement, total duration, and predictors. J Rheumatol. 2014 Jun;41(6):1163-70. doi: 10.3899/jrheum.131503. Epub 2014 May 1. PMID 24786928
- [Derived] Wallace CA, Giannini EH, Spalding SJ, Hashkes PJ, O'Neil KM, Zeft AS, Szer IS, Ringold S, Brunner HI, Schanberg LE, Sundel RP, Milojevic D, Punaro MG, Chira P, Gottlieb BS, Higgins GC, Ilowite NT, Kimura Y, Hamilton S, Johnson A, Huang B, Lovell DJ; Childhood Arthritis and Rheumatology Research Alliance. Trial of early aggressive therapy in polyarticular juvenile idiopathic arthritis. Arthritis Rheum. 2012 Jun;64(6):2012-21. doi: 10.1002/art.34343. Epub 2011 Dec 19. PMID 22183975
- See also: Click here for the Childhood Arthritis and Rheumatology Research Alliance (CARRA) Web site — http://www.carragroup.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 children with poly JIA within 12 months of onset recruited from pediatric rheumatology clinics at 15 sites
Pre-assignment Details: Eligible patients were permitted to have received up to 2 intra-articular corticosteroid injections before or up to 2 weeks after baseline; and oral prednisolone for up to 4 weeks, but must have been off corticosteroids for at least 1 week prior to enrollment. Patients with past or current JIA-associated uveitis were excluded.
Groups:
- Methotrexate-Prednisolone-Etanercept Arm: Methotrexate 0.5 mg/kg given by subcutaneous injection once per week, plus etanercept 0.8 mg/kg given by subcutaneous injection once per week, plus prednisolone by mouth daily with decreasing dose tapered over 16 weeks
Period: Overall Study
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm
Started | 43 | 42
Completed | 39 | 38
Not Completed | 4 | 4
Not completed — Lack of Efficacy | 3 | 3
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 patients were ineligible
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 42 | 85
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.1 (4.1) | 9.9 (4.6) | 10.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 9 | 13 | 22
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Attain Inactive Disease by 6 Months
Time Frame: 6 months after initiation of study intervention
Population: all participants receiving study medications
Measure: Number; unit: participants
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm
Number analyzed (Participants) | 43 | 42
participants | 10 | 17

2. Secondary Outcome: Safety Profiles, Including the Number of Treatment-emergent, Serious, or Unexpected Adverse Events and Other Important Medical Events
Time Frame: Over 12 months maximum study participation per subject
Population: all participants that received study medications
Measure: Number; unit: events
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm
Number analyzed (Participants) | 43 | 42
events | 1 | 2

3. Secondary Outcome: Clinical Remission on Medication
Description: 6 months of clinical inactive disease
Time Frame: 12 months or end of study
Population: all participants receiving study medications
Measure: Number; unit: participants
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm
Number analyzed (Participants) | 43 | 42
participants | 3 | 9

ADVERSE EVENTS:
Arm/Group | Methotrexate Arm | Methotrexate-Prednisolone-Etanercept Arm
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/42
Other Adverse Events (participants affected / at risk) | 0/43 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate Arm (N=43) | Methotrexate-Prednisolone-Etanercept Arm (N=42)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — This participant withdrew from the study, the event resolved without sequelae
psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — Participant on open label medications had acute psyhotic event that resolved with tapering of prednisolone. Patient continued in the study.
septic hip (Infections and infestations) | 0 (0) | 1 (1) — after discontinuation of open label therapy for 2 months, patient was found to have infection of the hip, this resolved. No organism was recovered.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate Arm (N=43) | Methotrexate-Prednisolone-Etanercept Arm (N=42)
liver function test elevation (Hepatobiliary disorders) | 0 (0) | 3 (3) — elevation of LFT grade 3

LIMITATIONS AND CAVEATS:
small number of participants with recent onset poly JIA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No